CLINICAL TRIAL: NCT03255837
Title: A Single Blind, Randomized Controlled Trial of Anodal Transcranial Direct-current Stimulation (tDCS) Against Cathodal and Sham Stimulation in Adults With High-Functioning Autism
Brief Title: tDCS on Working Memory (WM) in Adults With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GN17MH365
Record Dates: First submitted 2017-08-16; First posted 2017-08-21 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Transcranial Stimulation; Memory
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Each participant will receive the same 3 kinds of transcranial stimulation. However, the order in which they receive them will be randomly allocated.
Who Masked: Participant
Masking Description: Participants will be unaware of the order in which they receive the transcranial stimulation condition (anodal, cathodal, sham).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcranial direct current stimulation (tDCS) - anodal (Experimental): Transcranial direct current stimulation - anodal (positive) 1.5 millamps for 15 minutes
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Transcranial direct current stimulation (tDCS) - cathodal (Experimental): Transcranial direct current stimulation - cathodal (negative) 1.5 millamps for 15 minutes
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Transcranial direct current stimulation (tDCS) - sham (Sham Comparator): Transcranial direct current stimulation - sham session 15 minutes
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Transcranial Direct Current Stimulation (tDCS, a form of non-invasive brain stimulation) on the left dorsolateral prefrontal cortex (DLPFC)

SUMMARY:
This study will involve an experiment in individuals with Autism Spectrum Disorder (ASD) comparing their performance on a working memory task before, during and after non-invasive brain stimulation (tDCS) compared to a control group in a 3x3 factorial design. How the stimulation affects performance on the task will be assessed, along with the impact of the intervention on the individuals.

DETAILED DESCRIPTION:
Many studies have examined working memory in people with autism spectrum disorder as working memory deficits in individuals with autism spectrum disorder leads to multiple difficulties associated with behaviour regulation, cognitive flexibility, abstract thinking, and focusing and sustaining attention. Evidence suggests that transcranial Direct Current Stimulation on the left dorsolateral prefrontal cortex leads to an increase in working memory performance in typically developing individuals. This may have important benefits for people with autism spectrum disorder since autism spectrum disorder is known to be associated with working memory deficiencies. This study will build on a pilot study conducted in 2014, the experiment tested participants working memory scores on an N-back test, after receiving anodal (positive stimulation) stimulation for 15 minutes over the left dorsolateral prefrontal cortex. This task requires the participant to perform multiple cognitive operations, including encoding of new stimuli, updating and maintaining past stimuli, and recognising and responding to whether each new stimulus matches the three-back stimulus. Participants are presented with a random set of ten letters (from A-Z). A different letter will be displayed every 2s, participants will be required to respond (key press 1) if the presented letter was the same as the letter presented three stimuli previously (a target). If it was not a target, participants were required to respond with key press 2. In this test, a total of 30 correct responses are possible. Participants will perform the task three times to reduce variability. Accuracy (number of correct responses), error rate (number of incorrect responses), and reaction time (interval between target presentation and pressing 1 or 2) will be recorded. Based on the findings from the pilot study, a full study will be conducted to investigate the effects of anodal transcranial Direct Current Stimulation on adults with high-functioning autism, as well as test whether the effects of transcranial Direct Current Stimulation on dorsolateral prefrontal cortex is dependent on polarity (anodal versus cathodal (negative stimulation) stimulation).

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of ASD
* right handed
* speaks English fluently
* normal vision or corrected to normal
* passing tDCS safety screening

Exclusion Criteria:

* participants who do not understand verbal or written English (i.e would be in need of translators)
* participants that have ever suffered from epilepsy, febrile convulsions in infancy or had recurrent fainting spells
* family history of epilepsy
* has a heart pacemaker, cochlear implant, medication pump, surgical clips
* has drunk more than 3 units of alcohol in the last 24 hours
* suffers from migraines
* metal in the head, implanted brain medical devices
* has undergone a neurosurgical procedure
* has had more than one cup of coffee, or other sources of caffeine in the last hour
* taking any unprescribed or prescribed medication that might effect tDCS
* medications or psychoactive drugs that can lower seizure threshold [imipramine, amitriptyline, doxepine, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine, (MDMA, ecstasy), phencyclidine (PCP, angel dust), ketamine, gamma-hydroxybutyrate (GHB), alcohol, theophylline]
* withdrawal from alcohol, barbiturates, benzodiazepines, meprobamate, chloral hydrate

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Working memory accuracy score compared to typically developed controls scores. | Change from baseline (before stimulation) to after stimulation (1 week)
  Result of N-back memory task

SECONDARY OUTCOMES:
Difference in working memory accuracy score between adults with ASD and healthy controls | Before stimulation
  Result of N-back memory task
Difference in working memory accuracy score between adults with ASD and healthy controls | After stimulation (1 week)
  Result of N-back memory task

CONTACTS AND LOCATIONS:
Overall Officials: Craig Melville, MD, Study Director — University of Glasgo
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No